CLINICAL TRIAL: NCT03190577
Title: Assessment of the Prevalence of TTR Amyloid Neuropathy in a Population of Patients With Neuropathy of Unknown Aetiology
Acronym: PRE-TRANS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC16_0427
Record Dates: First submitted 2017-06-14; First posted 2017-06-19 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Familial Amyloid Neuropathy; Transthyretin Amyloidosis
Keywords: Transthyretin mutation
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Amyloidosis, Hereditary, Transthyretin-Related | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with neuropathy of unknown aetiology (Experimental): from a blood sample performed at inclusion, a genetic analysis will be performed to research transthyretin mutation
  Interventions: Genetic: blood sample

INTERVENTIONS:
Genetic: blood sample — two 5 ML EDTA tubes of blood will be collected once by patient

SUMMARY:
Familial amyloid neuropathy due to transthyretin gene mutations (TTR-FAP) is a rare autosomal dominant inherited disease resulting in the abnormal multi-system deposition of amyloid proteins. These deposits produce a multi-organ disease. AP is usually fatal 10 to 15 years after onset of symptoms if untreated. The prevalence of the disease remains still poorly understood and usually the search for this pathology is done in a third line of investigation. So the average time to diagnosis is extremely long, from 12 to 24 month. Now that the investigators have etiological treatment ( famidis (Vyndaqel®) and Diflunisal (Dolobid)) of this disease, it is essential to be able to detect FAP patients as early as possible. With this study, investigator decided to test for TTR mutation all patients presented with neuropathy of unknown etiology at the first line of investigation. The goal of this study is to evaluate the prevalence of FAP-TTR among neuropathy and defined the best strategy to test this population for TTR mutations.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (male and female) aged not more than 90 years old
* Patients with neuropathy identified by EDX exam or small fibre neuropathy identified from a skin biopsy.
* Patients who have undergone the minimal assessment for neuropathy as defined by the HAS (French National Health Authority): biological analysis (fasting glucose, CBC, liver and renal functions, CRP, pituitary TSH)
* Patients belonging to the social security system
* Patient who gave written informed consent

NON-INCLUSION CRITERIA Patients under legal supervision or guardianship Patients with a confirmed documented diagnosis of the cause of neuropathy Patients with evidence of Charcot Marie Tooth neuropathy: very slowly progressive course, pes cavus.

Patients who have already been investigated for a TTR mutation Pregnant women Minors

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
to evaluate the prevalence of TTR amyloidosis | inclusion
  number of patients with TTR mutation

SECONDARY OUTCOMES:
To identify risk factors of carrying TTR mutations amongst those presenting with "unknown aetiology" neuropathy | inclusion
  comparison between patient of medical history, alcohol use, familial neuropathy history, age of first symptoms apparition, description of first symptoms
Description of the TTR-FAP cohort | inclusion
  medical history, alcohol use, smoking habits, familial neuropathy history, age of first symptoms apparition, description of first symptoms

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - Chu Angers, Angers
  - Chru Brest, Brest
  - Chd La Roche Sur Yon, La Roche-sur-Yon
  - Ch La Rochelle, La Rochelle
  - Ch Le Mans, Le Mans
  - Chu Nantes, Nantes
  - Chu Poitiers, Poitiers
  - Ch Quimper, Quimper
  - Ch Saint Brieuc, Saint-Brieuc
  - CHP Saint-Grégoire - Cabinet de Neurologie ENMG, Saint-Grégoire
  - Ch Saint Nazaire, Saint-Nazaire
  - Chru Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Magot A, Lepetit M, Genestet S, Noury JB, Ollivier Y, Lejeune P, Metzger L, Beltran S, Cassereau J, Pihan M, Kolev I, Pegat B, Boyer K, Stancu A, Baron C, Dahimene F, Perrault C, Martineau AS, Pere M, Bezieau S, Kyndt F, Pereon Y. Etiologic Diagnosis of Neuropathies Based on First-Line Screening of TTR Gene Mutations. J Peripher Nerv Syst. 2025 Sep;30(3):e70043. doi: 10.1111/jns.70043. PMID 40586114